CLINICAL TRIAL: NCT05408702
Title: Barriers and Facilitators to Exercise for Individuals With Autoimmune Myasthenia Gravis, Congenital Myasthenic Syndrome or Lambert-Eaton Myasthenic Syndrome in France: a Descriptive, Cross-sectional Study
Brief Title: Exercise in Autoimmune Myasthenia Gravis and Myasthenic Syndromes
Acronym: MYaEX
Status: Completed | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Principal Investigator, Simone BIRNBAUM, Principal Investigator, Institut de Myologie, France
Other Study IDs: MYaEX
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Autoimmune Myasthenia Gravis; Lambert-Eaton Myasthenic Syndrome; Congenital Myasthenic Syndrome; Myasthenia Gravis
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome; Myasthenic Syndromes, Congenital; Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Autoimmune Myasthenia Gravis
- Congenital Myasthenic Syndrome
- Lambert Eaton Syndrome

SUMMARY:
A few recent observational studies show that despite the lack of clear recommendations, many individuals with myasthenia participate in exercise. However, no link has been found between exercise and the severity of myasthenia symptoms, measured by the Muscle Myasthenia Score or the Myasthenia Gravis Composite Score. This suggests that there are other factors that may limit or prevent some individuals from being active, or factors which may facilitate participation in exercise.

Studies in other diseases have shown that there are internal (beliefs, motivation, etc.) and external (cost, accessibility, etc.) factors unrelated to the disease which may play a role in exercise participation.

The aim of this study is to identify factors that facilitate or limit exercise in individuals with autoimmune myasthenia gravis, congenital myasthenia syndrome and Lambert-Eaton syndrome.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* confirmed diagnosis of MG or SMC or LEMS
* Live in France or its territories
* Provide consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living in France or its territories, with a confirmed diagnosis of MG or SMC or LEMS
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Barriers and facilitators to exercise | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Online Questionnaire, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided